CLINICAL TRIAL: NCT05260671
Title: An Exploratory Clinical Study to Evaluate the Efficacy and Safety of Penpulimab in Combination With Cetuximab as First-line Treatment in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (R/MSCCHN)
Brief Title: Penpulimab in Combination With Cetuximab as First-line Treatment in R/M SCCHN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Wang Xiaoshen, director, Eye & ENT Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-C-SCCHN
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Neoplasms; Recurrent Disease; Metastatic Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penpulimab+cetuximab (Experimental): Erbitux 500 mg/m2 without immunotherapy for 14 days prior to the first cycle. Cetuximab Injection 500 mg/m2 and Penpulimab Injection 200 mg are intravenously infused on Day 1 (D1) of Cycle 1, with 14 days as one cycle. Penpulimab for up to 96 weeks (48 cycles)
  Interventions: Drug: Penpulimab combined with cetuximab

INTERVENTIONS:
Drug: Penpulimab combined with cetuximab — PD-1 antibody combined with EGFR inhibitors, biweekly
  Other Names: AK105+Erbitux

SUMMARY:
This trial is a multicenter, prospective, single-arm exploratory clinical study to evaluate the efficacy and safety of Penpulimab injection combined with cetuximab in the first-line treatment of recurrent/metastatic squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
Based on the apparent efficacy and favorable safety profile of previous PD-1 and cetuximab combination therapy, Penpulimab (PD-1 antibody) combined with cetuximab in the first-line treatment of patients with recurrent/metastatic SCCHN are used to assess the efficacy and safety of the regimen. Among them, Penpulimab (PD-1 antibody) is approved for adult patients with relapsed or refractory classical Hodgkin's lymphoma who have received at least second-line systemic chemotherapy in China. Cetuximab is approved in China for first-line treatment of recurrent/metastatic SCCHN in combination with chemotherapeutic drugs platinum and fluorouracil.

This study plans to enroll 48 patients with untreated recurrent/metastatic squamous cell carcinoma of the head and neck who will receive Penpulimab injection combined with cetuximab. Cetuximab 500 mg/m2 without PD-1 drugs for 14 days prior to Cycle 1. Cetuximab Injection 500 mg/m2 and Penpulimab Injection 200 mg are intravenously infused on Day 1 (D1) of Cycle 1, with 2 weeks (14 days) as a cycle. Penpulimab will be administered for no more than 96 weeks (48 cycles), and cetuximab will be administered until disease progression, unacceptable toxicity, or withdrawal decision by the subject.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years, male or female;
* Histologically confirmed squamous cell carcinoma of the head and neck (oral cavity, oropharynx, larynx, hypopharynx) (SCCHN);
* Recurrent/metastatic SCCHN not suitable for local treatment such as surgery or radiotherapy in the opinion of the investigator;
* At least one measurable tumor lesion according to RECIST 1.1 criteria;
* The tumor expresses PD-L1, with a comprehensive positive score CPS ≥ 1;
* Eastern Cooperative Oncology Group (ECOG) PS: 0-1
* Expected survival ≥ 3 months;
* Normal function of major organs, meeting the following criteria: blood routine examination criteria must be met: (no blood transfusion within 14 days before screening) 1) HB ≥ 90 g/L; 2) ANC ≥ 1.5 × 109/L; 3) PLT ≥ 75 × 109/L; biochemistry: (without transfusion or blood product within 14 days before screening) 1) BIL ≤ 1.5 × upper limit of normal (ULN) (≤ 3 × ULN for patients with Gilbert's syndrome); 2) ALT and AST ≤ 2.5 × ULN (≤ 5 × ULN for patients with liver metastasis); 3) Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50ml/min (Cockcroft-Gault formula); 4) Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN; left ventricular ejection fraction (LVEF) ≥ 50% assessed by cardiac Doppler ultrasound;
* Women of childbearing potential must have a negative pregnancy test (serum or urine) within 14 days prior to enrollment and are willing to use reliable contraception during the trial and must be non-lactating patients; male subjects must use reliable contraception from the start of treatment to 6 months after the last dose;
* The subjects voluntarily join the study, sign the ICF, have good compliance, and cooperate in the follow-up

Exclusion Criteria:

* Received systemic chemotherapy, but excluding chemotherapy for locally advanced disease as a part of multimodal treatment. Note: Chemotherapy for locally advanced disease includes induction chemotherapy, radiotherapy with concurrent chemotherapy, and adjuvant chemotherapy;
* Previous immunotherapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibodies or any other antibody or drug specifically targeting T cell costimulation or immune checkpoint pathways;
* Previous use of anti-EGFR drugs such as cetuximab, nimotuzumab, gefitinib, and afatinib;
* Pregnant or lactating, or planning to become pregnant during the study period;
* Current participation and receipt of study treatment, or participation in an investigational drug trial or use of an investigational device within 4 weeks prior to randomization;
* Presence of uncontrolled or symptomatic active central nervous system (CNS) metastases, which may present with clinical symptoms, cerebral edema, spinal cord compression, carcinomatous meningitis, leptomeningeal disease, and/or progressive growth;
* Any active autoimmune disease or history of autoimmune disease (but not limited to autoimmune hepatitis, interstitial pneumonia, enteritis, hypophysitis, vasculitis, nephritis; positive HIV test or history of the above diseases, or history of organ transplantation; but the following patients are allowed: vitiligo, psoriasis, alopecia, well-controlled type I diabetes mellitus, Hypothyroidism with euthyroidism treated by replacement therapy;
* Treatment with systemic immunosuppressive drugs within 2 weeks before the start of study treatment or anticipation of the need for systemic immunosuppressive drugs during study treatment, with the following exceptions: 1) Intranasal, inhaled, topical steroids, or topical steroids (e.g., intra-articular); 2) Physiological doses of systemic corticosteroids (≤ 10 mg/day prednisone or equivalent); 3) Steroid premedication for hypersensitivity (e.g., premedication for CT scan);
* Significant cardiovascular disease, such as cardiac insufficiency above class II (New York Heart Association (NYHA) classification) or left ventricular ejection fraction < 50%, unstable angina pectoris, myocardial infarction within 1 year, arrhythmia requiring treatment, QTc ≥ 450 ms (male), QTc ≥ 470 ms (female);
* The subject has an active infection or infectious disease, requiring systemic antibacterial, antifungal, or antiviral treatment, including tuberculosis infection; or has an unexplained fever (body temperature > 38.5℃) during the screening period or prior to the first dose;
* Interstitial lung disease or non-infectious lung disease (including past medical history and prevalence), uncontrolled systemic diseases, including pulmonary fibrosis, acute lung disease, diabetes (fasting blood glucose (FBG) > 8.9 mmol/L), hypertension (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 90 mmHg), kidney disease (urine routine showed urine protein ≥ 2 +, or 24 h urine protein quantification > 1.0g), etc., except for local interstitial pneumonia induced by radiotherapy;
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
* Subjects with a history of other malignancies within the past 5 years, but except for cured cervical carcinoma in situ, squamous cell carcinoma of the skin, basal cell carcinoma of the skin, localized prostate cancer, or other carcinomas in situ with definitive resection;
* Virological screening meets any of the following criteria: hepatitis B HBsAg positive and HBV-DNA ≥ 10^3 copies/ml; hepatitis C: HCV antibody positive and HCV-RNA positive (results greater than the lower limit of detection of the analytical method);
* Participants may need to be vaccinated during the study or have received a live viral vaccine within 4 weeks prior to enrollment. Seasonal influenza vaccine without live virus is permitted.
* Patients with other concomitant diseases that seriously jeopardize the patient's safety or affect the patient's completion of the study, as judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2 years
  Defined as the percentage of complete response (CR) or partial response (PR) (i.e., CR + PR) evaluated according to RECIST v1.1 from the start of trial medication

SECONDARY OUTCOMES:
Overall survival | 2 years
  Time from start of trial medication to death due to any cause.
Progression-free survival | 2 years
  Defined as the time from the start of trial medication to either PD as assessed by RECIST v 1.1 or death due to any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoshen Wang, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (2):
- China (2):
  - Department of radiotherapy,The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Department of Radiotherapy, Eye & ENT Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No